CLINICAL TRIAL: NCT02995720
Title: An Open-label, Randomized, Single-dose, 2X3X3 Partial Replicate, Crossover Study to Compare the Pharmacokinetics and Safety Between a Fixed Dose Combination of Fimasartan/Amlodipine/Rosuvastatin and Co-administration of a Fixed Dose Combination of Fimasartan/Amlodipine and Rosuvastatin in Healthy Male Subjects
Brief Title: A Study to Compare the Pharmacokinetics and Safety of a Fixed Dose Combination of Fimasartan/Amlodipine/Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FARC-CT-103
Record Dates: First submitted 2016-12-01; First posted 2016-12-16 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Hypertension, Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — fimasartan; Rosuvastatin Calcium

ARMS (2):
- 1 (Experimental): A fixed dose combination of Fimasartan/Amlodipine/Rosuvastatin
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Rosuvastatin
- 2 (Active Comparator): Co-administration of Fimasartan/Amlodipine combination drug and Rosuvastatin
  Interventions: Drug: Fimasartan/Amlodipine combination drug, Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan/Amlodipine combination drug, Rosuvastatin

SUMMARY:
An open-label, randomized, single-dose, 2X3X3 partial replicate, crossover study to compare the pharmacokinetics and safety between a fixed dose combination of Fimasartan/Amlodipine/Rosuvastatin and Co-administration of a fixed dose combination of Fimasartan/Amlodipine and Rosuvastatin in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject, aged 19- 50 years

Exclusion Criteria:

* History of clinically significant hypersensitivity to study drug, any other drug
* Hypotension or hypertension
* Active liver disease
* History of gastrointestinal disease
* History of excessive alcohol abuse
* Participation in any other study within 3 months

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum concentration of drug in plasma) of Fimasartan, Amlodipine and Rosuvastatin | 0~72 hour after medication
AUCt (Area Under the Curve from the dosing time to the last measurable concentration) of Fimasartan, Amlodipine and Rosuvastatin | 0~72 hour after medication